CLINICAL TRIAL: NCT06116682
Title: A Phase II Study of Amivantamab SC (Subcutaneous) in Participants With MET Amplification-Positive Stage IV or Recurrent Non-Small Cell Lung Cancer (LUNG-MAP SUB-STUDY)
Brief Title: Targeted Treatment for Advanced Non-Small Cell Lung Cancer That Has Increased Copies of the MET Gene (An Expanded Lung-MAP Treatment Trial)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S1900J; NCI-2023-07072 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1900J (Other: SWOG); S1900J (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Lung Non-Small Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — amivantamab; Specimen Handling; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (amivantamab) (Experimental): Patients receive amivantamab SC on days 1, 8, 15, and 22 of cycle 1 and then on days 1 and 15 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI and collection of blood samples throughout the trial.
  Interventions: Biological: Amivantamab; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Biological: Amivantamab — Given amivantamab-SC
  Other Names: Amivantamab-vmjw; Anti-EGFR/c-Met Bispecific Antibody JNJ-61186372; CNTO-4424; JNJ 61186372; JNJ-611; JNJ-61186372; JNJ61186372; Rybrevant
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI

SUMMARY:
This phase II Expanded Lung-MAP treatment trial tests how well amivantamab-subcutaneous (SC) works in treating patients patients with MET amplification non-small cell lung cancer. Amivantamab-SC is a drug that reduces extra copies of the MET gene, a change present in your tumor. Giving amivantamab-SC may lower the chance of the growth or spread of advanced non-small cell lung cancer that has extra copies of the MET gene in the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the objective response rate (ORR) (confirmed and unconfirmed, complete and partial) in participants with MET amplification-positive non-small cell lung cancer (NSCLC) treated with amivantamab-SC within each cohort.

SECONDARY OBJECTIVES:

I. To evaluate progression-free survival (PFS) within each cohort. II. To evaluate overall survival (OS) within each cohort. III. To evaluate the duration of response among responders within each cohort. IV. To evaluate the frequency and severity of toxicities within each cohort and combined across all study participants.

TRANSLATIONAL MEDICINE OBJECTIVES:

I. To collect, process, and bank cell-free deoxyribonucleic acid (cfDNA) prior to treatment on Cycle 1 Day 1, Cycle 3 Day 1, and at first progression for future development of a proposal to evaluate comprehensive next-generation sequencing of circulating tumor deoxyribonucleic acid (ctDNA).

II. To establish a tissue/blood repository from participants with refractory non-small cell lung cancer (NSCLC).

OUTLINE:

Patients receive amivantamab subcutaneously (SC) on days 1, 8, 15, and 22 of cycle 1 and then on days 1 and 15 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo computerized tomography (CT) or magnetic resonance imaging (MRI) and collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have been assigned to S1900J by the Southwest Oncology Group (SWOG) Statistics and Data Management Center (SDMC). Assignment to S1900J is determined by the LUNGMAP protocol
* Participants must have documentation of NSCLC with MET amplification determined by FMI tissue-based next generation sequencing (NGS) assay
* Participants must have measurable disease documented by CT or MRI. The CT from a combined positron emission tomography (PET)/CT may be used to document measurable disease ONLY if it is of diagnostic quality: otherwise, it may be used to document non-measurable disease only. Measurable disease must be assessed within 28 days prior to sub-study registration. Pleural effusions, ascites and laboratory parameters are not acceptable as the only evidence of disease. Non-measurable disease must be assessed within 42 days prior to sub-study registration. All known sites of disease must be assessed and documented on the Baseline Tumor Assessment Form. Participants whose only measurable disease is within a previous radiation therapy port must demonstrate clearly progressive disease (in the opinion of the treating investigator) prior to sub-study registration to be considered measurable
* Participants must have a CT or MRI scan of the brain to evaluate for central nervous system (CNS) disease within 42 days prior to sub-study registration
* Participants with asymptomatic CNS metastasis (brain metastases or leptomeningeal disease) must be clinically stable and asymptomatic for at least 14 days prior to sub-study registration

  * NOTE: Participants can be on a low-dose corticosteroid treatment (≤ 10 mg prednisone or equivalent) for at least 14 days prior to study treatment
* Participants must not have other known actionable oncogenic alterations, such as (but not limited to) EGFR sensitizing mutations, EGFR T790M mutation, MET Exon-14 skipping mutant NSCLC, ALK gene fusion, ROS1 gene rearrangement, RET gene rearrangement, NTRK rearrangement, HER2 mutation, KRAS activating mutations, and BRAF V600E mutation
* Participants must have progressed (in the opinion of the treating physician) following the most recent line of therapy
* Participants must have received at least one line of systemic treatment for Stage IV or recurrent NSCLC
* Participants must have recovered (≤ Grade 1) from any side effects of prior therapy. The exception is if a side effect from a prior treatment is known to be permanent without expected further recovery or resolution (i.e., endocrinopathy from immunotherapy or cisplatin neurotoxicity)
* Participants must not have been previously treated for any cancer with MET tyrosine kinase inhibitors (TKIs) such as tepotinib, capmatinib, and crizotinib
* Participants must not have received any prior systemic therapy (systemic chemotherapy, immunotherapy or investigational drug) within 21 days prior to sub-study registration
* Participants must not have a prior treatment with anti-PD-1 or anti-PD-L1 antibody within 6 weeks of sub-study registration
* Participants must not have received any radiation therapy within 14 days prior to sub-study registration
* Participants must not be planning to receive any concurrent chemotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment while receiving treatment on this study
* Participants must not have had major surgery excluding placement of vascular access or tumor biopsy, or had significant traumatic injury within 28 days prior to sub-study registration, or will not have fully recovered from surgery, or has surgery planned during the time the participant is expected to participate in the study

  * NOTE: Participants with planned surgical procedures to be conducted under local anesthesia may participate
* Participants must not have a prior or concurrent malignancy whose natural history or treatment (in the opinion of the treating physician) has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Absolute neutrophil count ≥ 1.5 x 10^3/uL (within 28 days prior to sub-study registration)
* Hemoglobin >= 10.0 g/dL (within 28 days prior to sub-study registration)
* Platelets ≥ 75 x 10^3/uL (within 28 days prior to sub-study registration)
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) unless history of Gilbert's disease. Participants with history of Gilbert's disease must have total bilirubin ≤ 5 x institutional ULN (within 28 days prior to sub-study registration)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × institutional ULN. Participants with history of liver metastasis must have AST and ALT ≤ 5 x ULN (within 28 days prior to sub-study registration)
* Participants must have a serum creatinine ≤ the institutional upper limit of normal (IULN) or calculated creatinine clearance ≥ 45 mL/min using the following Cockcroft-Gault Formula. This specimen must have been drawn and processed within 28 days prior to sub-study registration. For creatinine clearance formula see the tools on the CRA Workbench
* Participants' most recent Zubrod performance status must be 0-2 and be documented within 28 days prior to sub-study registration
* Participants must have a completed medical history and physical exam within 28 days prior to sub-study registration
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, must have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants must be class 2B or better
* Participants with known human immunodeficiency virus (HIV)-infection must be on effective anti-retroviral therapy and have undetectable viral load test on the most recent test results obtained within 6 months prior to sub-study registration
* Participants with evidence of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load while on suppressive therapy on the most recent test results obtained within 6 months prior to sub-study registration
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. Participants currently being treated for HCV infection must have undetectable HCV viral load test on the most recent test results obtained within 6 months prior to sub-study registration
* Participants with known diabetes as determined by the treating investigator must show evidence of controlled disease within 14 days prior to sub-study registration
* Participants of reproductive potential must have a negative serum pregnancy test within 7 days prior to sub-study registration
* Participants must not have other clinically active infectious liver disease
* Participants must not have clinically significant hypertension within 28 days prior to sub-study registration as determined by the treating investigator
* Participants must not have a history of pneumonitis that required drug therapy or an active symptomatic interstitial lung disease (ILD)/pneumonitis, including drug-induced or radiation ILD/pneumonitis
* Participants must not have ongoing or active infection or be diagnosed or suspected viral infection as determined by the treating investigator. NOTE: Participants that have an infection requiring antimicrobial therapy will be required to complete antibiotics 1 week prior to starting treatment
* Participants must not have active bleeding diathesis as determined by the treating investigator
* Participants must not have impaired oxygenation requiring continuous oxygen supplementation as determined by the treating investigator
* Participants must not have psychiatric illness, social situation, or any other circumstances that would limit compliance with study requirements as determined by the treating investigator
* Participants must not have any ophthalmologic condition that is unstable in the opinion of the treating investigator
* Participants must not be pregnant or breastfeeding (nursing includes breast milk fed to an infant by any means, including from the breast, milk expressed by hand, or pumped). Individuals who are of reproductive potential must have agreed to use an effective contraceptive method with details provided as a part of the consent process. A person who has had menses at any time in the preceding 12 consecutive months or who has semen likely to contain sperm is considered to be of "reproductive potential." In addition to routine contraceptive methods, "effective contraception" also includes refraining from sexual activity that might result in pregnancy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) including hysterectomy, bilateral oophorectomy, bilateral tubal ligation/occlusion, and vasectomy with testing showing no sperm in the semen
* Participants must agree to have blood specimens submitted for circulating tumor DNA (ctDNA)
* Participants must also be offered participation in specimen banking. With participant consent, specimens must be collected and submitted via the SWOG Specimen Tracking System
* Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines

  * NOTE: Participants with impaired decision-making capabilities, legally authorized representatives may sign and give informed consent on behalf of study participants in accordance with applicable federal, local, and Central Institutional Review Board (CIRB) regulations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Response rate for amivantamab-subcutaneous | Up to 3 years
  Response rates and associated confidence intervals will be calculated.

SECONDARY OUTCOMES:
Overall survival | Up to 3 years
  Will be estimated using the method of Kaplan-Meier. The Brookmeyer-Crowley method will be used to calculate confidence intervals for median times.
Progression free survival | Up to 3 years
  Will be estimated using the method of Kaplan-Meier. The Brookmeyer-Crowley method will be used to calculate confidence intervals for median times.
Duration of response | Up to 3 years
  Will be estimated using the method of Kaplan-Meier. The Brookmeyer-Crowley method will be used to calculate confidence intervals for median times.
Incidence of adverse events | Up to 28 days
  Toxicity will be evaluated among all participants enrolled on the study (combining the squamous and non-squamous cohorts). With 80 participants, any toxicity can be estimated to within 11% with 95% confidence. Any toxicity with at least 5% prevalence has at least a 98% chance of being observed.

CONTACTS AND LOCATIONS:
Overall Officials: Shirish Gadgeel, Principal Investigator — SWOG Cancer Research Network
Locations (213):
- United States (213):
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Sutter Auburn Faith Hospital, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Mills Health Center, San Mateo, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Bayhealth Hospital Sussex Campus, Milford, Delaware
  - Malcom Randall Veterans Administration Medical Center, Gainesville, Florida
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Advocate Outpatient Center - Aurora, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Advocate Outpatient Center - Oak Lawn, Oak Lawn, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate High Tech Medical Park, Palos Heights, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Virtua Samson Cancer Center, Moorestown, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - WellSpan Medical Oncology and Hematology, Chambersburg, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Cancer Center Dickson City, Dickson City, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - Ralph H Johnson VA Medical Center, Charleston, South Carolina
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin